CLINICAL TRIAL: NCT07049731
Title: Improvement of Skeletal and Muscle Health in Patients With Sarcopenia by AIBEN YUEDONG Protein Nutrition Powder in Combination With a Resistance Exercise Intervention
Brief Title: Improvement of Skeletal and Muscle Health in Patients With Sarcopenia by Protein Powder With Resistance Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weiwei Ma (Other)
Collaborators: Beijing Jishuitan Hospital, Capital Medical University (Unknown); Capital Medical University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Weiwei Ma, professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Z2025SY021
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo control group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo control
- Protein powder intervention group (Experimental)
  Interventions: Dietary Supplement: Protein powder intervention
- Resistance exercise+placebo control group (Experimental)
  Interventions: Behavioral: Resistance exercise intervention; Dietary Supplement: Placebo control
- Resistance exercise + protein powder intervention group (Experimental)
  Interventions: Dietary Supplement: Protein powder intervention; Behavioral: Resistance exercise intervention

INTERVENTIONS:
Dietary Supplement: Protein powder intervention — On the basis of a balanced diet, 2 sachets of Aiben Leap Protein Nutritional Powder (each sachet containing 6g of milk protein) were supplemented daily.
  Arms: Protein powder intervention group; Resistance exercise + protein powder intervention group
Behavioral: Resistance exercise intervention — Low-intensity resistance training was conducted 3 times a week.
  Arms: Resistance exercise + protein powder intervention group; Resistance exercise+placebo control group
Dietary Supplement: Placebo control — placebo was given and an individualized balanced dietary plan based on the Dietary Guidelines for Chinese Residents was provided.
  Arms: Placebo control group; Resistance exercise+placebo control group

SUMMARY:
Sarcopenia is an age-related progressive skeletal muscle disease, the prevalence of which is increasing year by year with the aging of China's population, seriously affecting the health and quality of life of the elderly. Relevant studies have shown that protein intake in combination with resistance exercise can significantly improve muscle mass and function, and the effect is superior to that of a single intervention. In addition, ingredients such as vitamin D, N-acetylglucosamine, sodium hyaluronate, and taurine can further promote muscle health by regulating metabolism and inflammation levels. However, there are relatively few intervention studies combining the above nutrients with resistance exercise in patients with sarcopenia. Therefore, this study intends to use protein powder containing milk protein, vitamin D, N-acetylglucosamine, sodium hyaluronate, taurine and other ingredients, combined with low-intensity resistance exercise, to intervene in the middle-aged and elderly patients with sarcopenia, and to explore and observe the effects on muscle mass, bone density, intestinal health and other indexes of patients with sarcopenia, with the aim of providing a more accurate nutritional and exercise intervention program for the prevention and treatment of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for sarcopenia AWGS 2019

  1. Grip strength less than 28.0 kg for males and less than 18.0 kg for females
  2. 6-meter stride speed less than 1.0 m/s or 5-repetition sit-up test time ≥ 12 seconds or SPPB ≤ 9 points.
  3. Bioelectrical Impedance Analysis (BIA) less than 7.0 kg/m² for males and 5.7 kg/m² for females or Dual-energy X-ray absorptiometry (DXA) less than 7.0 kg/m² for males and 5.4 kg/m² for females;
* Age between 35-75 years old with high compliance;
* Complete clinical data;
* Voluntary participation in the program with informed consent and signing of the informed consent form.

Exclusion Criteria:

* A clear history of allergy to protein powder in the past 6 months, or the presence of diarrhea symptoms and the frequency of ≥ 7 days / month, the duration of more than 2 weeks;
* Major physical diseases (diabetes with serious complications, malignant tumors, serious cardiovascular disease, neurological diseases or other diseases that may affect the effectiveness of exercise and nutritional interventions, etc.);
* The past three months, new fractures and recently underwent joint replacement surgery patients;
* Suffering from congenital bone or muscle diseases;
* The simultaneous existence of other comorbidities affecting muscle metabolism, such as malignant tumors, liver disease, severe organ insufficiency such as nephrotic syndrome, renal failure and other diseases that may affect protein metabolism;
* Participating in other clinical trials patients;
* With sensory disabilities or other reasons significantly affecting the collection of data, such as severe deafness, blindness, mental disorders, etc.;
* The researchers The researchers believe that other reasons are not suitable for clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Extremity Skeletal Muscle Mass Index (ASMI) | Baseline, month 3, month 6
  ASM was measured using BIA, ASMI=ASM/height (m)^2.
Handgrip strength | Baseline, month 3, month 6
  Maximum force grip was held for 3 seconds, the right and left hands were measured alternately, 3 measurements were taken in each hand, and the maximum value was taken.
6m walking speed | Baseline, month 3, month 6
  Let the tester start from the starting point, walk 6 meters at normal walking speed, stop when reaching the end point, record the time used, and calculate the 6m walking speed according to the time used and the distance of 6 meters.
Chair sitting and standing test | Baseline, month 3, month 6
  The subject sat in the center of the chair, crossed his/her arms in front of his/her chest, and after hearing the command "start", he/she completed 5 consecutive times of standing up and sitting down, and recorded the total time in seconds.
Simple Physical Performance Battery (SPPB) | Baseline, month 3, month 6
  The SPPB consists of 3 test items, each item is scored out of 4 points, and the total score is 12.

SECONDARY OUTCOMES:
General survey | Baseline, month 6
  Using a questionnaire designed by the research team and validated by the previous study, the survey covered the age, gender, ethnicity, marital status, occupation, education level, place of residence, household income, living status (living alone and with family), dietary habits and application of nutritional supplements, lifestyle (smoking, drinking, and physical activity), family history, and chronic diseases (hypertension, diabetes, etc.) of the study participants, Hyperlipidemia, etc.)
Height | Baseline, month 3, month 6
  Measure the height of the subjects
Weight | Baseline, month 3, month 6
  Measure the weight of the subjects
Body Mass Index(BMI) | Baseline, month 6
  Calculate BMI using height and weight , BMI=weight/(height)^2
Waist circumference, hip circumference, and waist to hip ratio | Baseline, month 3, month 6
  Measure the waist and hip circumference of the subjects and calculate the waist to hip ratio (waist circumference/hip circumference).
Body composition | Baseline, month 6
  Using a human body composition analyzer to detect indicators such as total score, visceral fat area, body segment fat and basal metabolic rate, body cell mass, and limb skeletal muscle mass index.
Assessment of ability to perform activities of daily living | Baseline, month 3, month 6
  The ADL was assessed using the Activity of Daily Living Scale (ADL), which consists of 10 items, including eating, bathing, grooming, dressing, bowel control, urination control, toileting, bed and chair transfers, walking, and walking up and down stairs.
  The total score is 100, with a score of more than 60 indicating mild functional impairment but basic self-care in daily life; a score of 60-41 indicating moderate functional impairment and need for some assistance in daily life; a score of 40-21 indicating severe functional impairment and obvious need for dependence on others in daily life; and a score of less than 20 indicating complete disability and total dependence on others in daily life.
Sleep assessment | Baseline, month 3, month 6
  The PSQI (Pittsburgh Sleep Quality Index) questionnaire was used to assess the quality of the subjects' sleep during the last 1 month. It consists of 19 self-assessment and 5 other-assessment entries, of which the 19th self-assessment and 5 other-assessment entries are not involved in scoring. The cumulative score of each component is the total PSQI score, which ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Analysis of dietary intake | Baseline, month 6
  The 3-day, 24-hour dietary recall method was used to investigate the subjects' dietary intake. The survey process was supplemented with tools such as the "Retrospective Dietary Survey Auxiliary Chart" to help the subjects accurately recall their dietary intake. Based on the Standardized Version of the Chinese Food Composition Table (6th Edition), the energy and various types of protein, fat and carbohydrate intake of the population were calculated, and for the missing data in the Chinese Food Composition Table, the United States Department of Agriculture Food Composition Table was used to supplement the data, so as to build up a comprehensive database of dietary intake. The analysis of dietary intake included the intake of total fat, total protein, total carbohydrates and energy and its percentage in the total energy intake.
Assessment of overall cognitive functioning | Baseline, month 6
  Subjects were assessed for overall cognitive functioning using the Montreal cognitive assessment (MoCA) scale out of 30, which contains cognitive functioning tests in multiple dimensions of visuospatial and executive functioning, naming, memory, attention, language, abstraction, delayed recall, and orientation.The normal threshold is usually ≥ 26 points, 21-25 points indicate mild cognitive impairment, and ≤ 20 points may indicate dementia risk
Bone density | Baseline, month 6
  Bone density, lumbar spine bone density (lumbar 2 - lumbar 4) and left femoral neck bone density are examined using the dualenergy X-ray absorptiometry (DXA) method.
Knee joint ultrasound | Baseline, month 6
  Ultrasound was used to examine the knee joint cavity for fluid or synovial hyperplasia and the tendon ligaments and muscles around the knee joint for damage.
Knee injury and osteoarthritis outcome score (KOOS score) | Baseline, month 3, month 6
  The KOOS rating includes five independent evaluation dimensions, each calculated separately and converted into a percentage scale (0-100 points, with higher scores indicating better functionality)
Serum sarcopenia related factors | Baseline, month 6
  Detect serum calcium (Ca), phosphorus (P), serum hydroxyvitamin D (25(OH)D), serum parathyroid hormone (PTH), P-alkaline phosphatase (ALP), serum osteocalcin (OC), serum type 1 pro-collagen N-terminal pre-peptide, serum type 1 collagen cross-linking N-terminal peptide (NTX), and serum anti-tartrate acid phosphatase 5b (TRACP-5b), estradiol (E2), leptin (LP), and so on.
Blood lipid concentration | Baseline, month 6
  Determine the serum levels of blood lipid concentration in the population. Lipid tests include total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C).
Blood glucose concentration | Baseline, month 6
  Blood glucose tests are fasting blood glucose.
Insulin concentration | Baseline, month 6
  Measurement of insulin secretion level.
Inflammation-related biochemical indicators | month 6
  Detecting inflammatory cytokine concentration: including TNF-α, IL-1 α, IL-1 β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-10 and other inflammatory factors.
Detection of intestinal flora species, quantity and differentiation level in human population | month 6
  The collected feces were subjected to 16S rRNA sequencing technology to detect the diversity of gut microbiota.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No